CLINICAL TRIAL: NCT03356340
Title: The Singapore Chinese Health Study
Acronym: SCHS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Woon-Puay Koh, Professor, National University of Singapore
Other Study IDs: SCHS
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Cancer; End Stage Renal Disease; Diabetes; Cardiovascular Diseases
MeSH Terms: conditions — Neoplasms; Kidney Failure, Chronic; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Beginning in April 1994, a 3% random sample of enrollees were re-contacted for donation of blood/buccal cells and spot urine specimens. In January 2001, the accrual of biospecimens was extended to include all consenting cohort enrollees. Hitherto, biospecimens have been collected from about 32,800 subjects (28,439 bloods, 4,438 buccal cells, 31,201 urines), representing a consent rate of about 60%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The "Singapore Chinese Health Study" is a cohort study established by the Department of Epidemiology and Public Health in National University of Singapore, together with collaborators from several universities in the United States of America. This is a long-term study to help doctors and scientists understand the influence of diet, lifestyle and environment on the development of common diseases among Singaporean men and women. This includes cancer, heart disease, stroke, dementia, osteoporosis, high cholesterol and diabetes. The aim is to help us understand the causes of these diseases and to discover effective and efficient approaches for prevention and treatment.

DETAILED DESCRIPTION:
The cohort consists of more than 60,000 men and women who were enrolled in the Singapore Chinese Health Study during 1993-1998. At the time of enrollment, participants were interviewed in-person regarding their dietary habits and other lifestyle factors. About half of them also donated small amounts of blood and urine for research between 2000 and 2004.

ELIGIBILITY:
Inclusion Criteria:

* Housing estate residents, ages 45-74 years, Chinese

Exclusion Criteria:

* None

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was established between April 1993 and December 1998 through the recruitment of a residential cohort of 63,257 Chinese men (n=27,959) and women (n=35,298), who were aged 45-74 years, and residing in public housing estates.
Sampling Method: Non-Probability Sample
Enrollment: 63257 (Actual)
Dates: Start 1993-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cancer incidence | 1993 to 2025
  Linkage to national cancer registry
End-stage Renal Disease | 1993 to 2025
  Linkage to national renal registry

REFERENCES:
- [Derived] Seah JYH, Ong CN, Koh WP, Yuan JM, van Dam RM. A Dietary Pattern Derived from Reduced Rank Regression and Fatty Acid Biomarkers Is Associated with Lower Risk of Type 2 Diabetes and Coronary Artery Disease in Chinese Adults. J Nutr. 2019 Nov 1;149(11):2001-2010. doi: 10.1093/jn/nxz164. PMID 31386157
- [Derived] Seah JYH, Koh WP, Yuan JM, van Dam RM. Rice intake and risk of type 2 diabetes: the Singapore Chinese Health Study. Eur J Nutr. 2019 Dec;58(8):3349-3360. doi: 10.1007/s00394-018-1879-7. Epub 2018 Dec 10. PMID 30535795
- [Derived] Lew QJ, Jafar TH, Jin A, Yuan JM, Koh WP. Consumption of Coffee but Not of Other Caffeine-Containing Beverages Reduces the Risk of End-Stage Renal Disease in the Singapore Chinese Health Study. J Nutr. 2018 Aug 1;148(8):1315-1322. doi: 10.1093/jn/nxy075. PMID 29986029
- [Derived] Neelakantan N, Koh WP, Yuan JM, van Dam RM. Diet-Quality Indexes Are Associated with a Lower Risk of Cardiovascular, Respiratory, and All-Cause Mortality among Chinese Adults. J Nutr. 2018 Aug 1;148(8):1323-1332. doi: 10.1093/jn/nxy094. PMID 29982724